

#### **OFFICIAL TITLE:**

A Phase 2, Randomized, Double-blind, Placebo-Controlled Efficacy, Pharmacokinetics and Safety Study of CA-008 in Subjects Undergoing Complete Abdominoplasty

# **NCT NUMBER:**

03789318

# **DOCUMENT DATE:**

24 April 2019



#### STATISTICAL ANALYSIS PLAN

# A Phase 2, Randomized, Double-blind, Placebo-Controlled Efficacy, Pharmacokinetics and Safety Study of CA-008 in Subjects Undergoing Complete Abdominoplasty

**Protocol Number: CA-PS-204** 

Protocol Version 2.0 (28JAN2019)

#### SPONSORED BY

Concentric Analgesics, Inc.

PREPARED BY
Lotus Clinical Research®, LLC
100 W California Blvd, Unit 25
Pasadena, CA 91105
626-397-2390 office
info@LotusCR.com
www.LotusCR.com

This document is confidential and proprietary to **Concentric Analgesics, Inc.** Acceptance of this document constitutes agreement by the recipient that no unpublished information contained herein will be reproduced, published, or otherwise disclosed without the prior written approval of **Concentric Analgesics, Inc.**, except that this document may be disclosed to appropriate Institutional Review Boards under the condition that they keep the information confidential.

Sponsor: Concentric Analgesics, Inc. Protocol Number: CA-PS-204

Statistical Analysis Plan Date: 24APR2019

# **DOCUMENT VERSION CONTROL**

| Version Number | Date | Comments/Changes |
|----------------|-----------|------------------|
| V1.0 | 24Apr2019 | SAP |


Sponsor: Concentric Analgesics, Inc. Protocol Number: CA-PS-204

Statistical Analysis Plan Date: 24APR2019

#### **APPROVALS**

Author:

DocuSigned by:

Napoleon Oleka

U

Signer Name: Napoleon Oleka

Signing Reason: I am the author of this document Signing Time: 4/28/2019 5:16:59 PM PDT

-F42C95E35B604F879437C6A49852CF9E

28-Apr-19

Date:

Napoleon Oleka

Senior Biostatistician

Lotus Clinical Research®, LLC

-DocuSigned by:

Jennifer Neyyer

Reviewed:

Approved:

Signer Name: Jennifer Nezzer

Signing Reason: I have reviewed this document Signing Time: 4/26/2019 8:34:33 PM PDT

F51546CD923C410C87CAB1F62D450C79

26-Apr-19

Date:

Jennifer Nezzer

Director, Biometrics

Lotus Clinical Research®, LLC

DocuSigned by:

Mike Royal

U

Signer Name: Mike Royal

Signing Reason: I approve this document Signing Time: 4/27/2019 12:43:03 PM PDT

608C20EC5FAD4832ADC799E971759505

27-Apr-19

Mike A. Royal, MD, JD, MBA

Chief Medical Officer

Concentric Analgesics Inc.

Date:


Statistical Analysis Plan Date: 24APR2019

# **TABLE OF CONTENTS**

| 1. | PURPOSE OF THE ANALYSES | 9 |
|-------|---------------------------------------------------|----|
| 2. | PROTOCOL SUMMARY | 9 |
| 2.1 | Study Objectives | 9 |
| 2.1.1 | Primary Objective | 9 |
| 2.1.2 | Secondary Objective | 9 |
| 2.2 | Overall Study Design and Plan | 9 |
| 2.2.1 | Study Stopping Rules | 11 |
| 2.2.2 | Study Population | 13 |
| 2.2.3 | Treatment Regimens | 13 |
| 2.2.4 | Treatment Group Assignments or Randomization | 13 |
| 2.2.5 | Sample Size Determination | 13 |
| 3. | GENERAL ANALYSIS AND REPORTING CONVENTIONS | 14 |
| 4. | SUBJECT POPULATIONS | 16 |
| 4.1 | Analysis Populations | 16 |
| 4.2 | Disposition of Subjects | 16 |
| 4.3 | Protocol Deviations | 17 |
| 5. | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | 17 |
| 5.1 | Demographics and Baseline Characteristics | 17 |
| 5.2 | Medical/Surgical History | 17 |
| 5.3 | Prior and Concomitant Medications | 17 |
| 6. | MEASUREMENTS OF TREATMENT EXPOSURE AND COMPLIANCE | 18 |
| 7. | EFFICACY EVALUATION | 19 |
| 7.1 | Handling of Dropouts or Missing Data | 19 |
| 7.2 | Sensitivity Analyses | 20 |
| 7.3 | Assessment Time Windows | 20 |
| 7.4 | Efficacy Endpoints | 21 |
| 7.4.1 | Primary Efficacy Endpoint | 21 |
| 7.4.2 | Key Secondary Efficacy Endpoints | 21 |

Sponsor: Concentric Analgesics, Inc. Protocol Number: CA-PS-204

Statistical Analysis Plan Date: 24APR2019

| 7.4.3 | Other Endpoints | .21 |
|---|---|---|
| 7.5 | Analysis Methods | .22 |
| 7.5.1 | NRS Measurements | .22 |
| 7.5.2 | Time-specific mean NRS pain intensity scores at T96h (Primary Efficacy Endpoint) and other time points | . 23 |
| 7.5.3 | AUC 0-96h at Rest (Key Secondary Efficacy Endpoint) and other AUC endpoint | nts23 |
| 7.5.4 | Time to opioid cessation or freedom (T <sub>OF</sub> ) (Key Secondary Efficacy Endpoint) | 23 |
| 7.5.5 | Opioid Free (OF) 24-96h (Key Secondary Efficacy Endpoint) and other timepoints. | . 24 |
| 7.5.6 | Total Opioid Consumption (OC) in Daily Oral Morphine equivalents 0-96h (Key Secondary Efficacy Endpoint) and other timepoints | |
| 7.5.7 | Percentage of Subjects who Rescue at T48 and other timepoints | 25 |
| 7.5.8 | PGE and IGE | .25 |
| 8. | SAFETY EVALUATION | .26 |
| 8.1 | Overview of Safety Analysis Methods | .26 |
| 8.2 | Adverse Events and SAEs | .26 |
| 8.3 | Physical Examination | .29 |
| 8.4 | Vital Signs | .30 |
| 8.5 | Surgical Site Assessments and Rebound (or Worsening) Pain Assessments | .30 |
| 8.6 | Neurosensory Test | .30 |
| 8.7 | ECG | . 31 |
| 8.8 | Clinical Laboratory Test Results | .31 |
| 8.9 | Drugs of Abuse and Alcohol Screens, Pregnancy Test | .31 |
| 8.10 | Subject Pain Assessment Training and Surgery Details | .31 |
| 9. | PHARMACOKINETIC EVALUATION | .31 |
| 10. | OTHER ANALYSES | . 32 |
| 11. | INTERIM ANALYSES | .32 |
| 12. | REFERENCES | .32 |
| 13. | APPENDICES | .32 |
| 13.1 | Planned Tables, Figures and Listings | .32 |
| 13.1.1 | Tables | .32 |
| 13.1.2 | Figures | . 35 |

Sponsor: Concentric Analgesics, Inc. Protocol Number: CA-PS-204

Statistical Analysis Plan Date: 24APR2019

| 13.1.3 | Listings | 36 |
|-----------|--------------------------------------------------------|----|
| 14. | DOCUMENT HISTORY | 37 |
| | LIST OF IN-TEXT TABLES AND FIGURES | |
| Table 2-1 | Protocol-Specified Visits and Visit Windows10 | ) |
| Table 2-2 | Study Stopping Rules | 2 |
| Table 3 | Equianalgesic Conversion Table25 | 5 |
| Table 4 | Table of Imputation Rules for Missing AE Start Dates29 | 9 |


#### LIST OF ABBREVIATIONS (COMMONLY USED)

ADaM Analysis Data Model

ADLs Actives of Daily Living

AE Adverse Event

ANOVA Analysis of variance

ATC Anatomical Therapeutic Chemical

AUC Area Under the Curve

BMI Body Mass Index

CDER Center for Drug Evaluation and Research

CP Completer

CRF Case Report Form

CRO Clinical Research Organization

CSR Clinical Study Report

ECG Electrocardiogram

EOS End of Study

ET Early Termination

FDA Food and Drug Administration

ICF Informed Consent Form

ICH International Conference on Harmonization

IGE Investigator Global Evaluation

ITT Intent-to-treat

LOCF Last Observation Carried Forward

MedDRA Medical Dictionary for Regulatory Activities

MED morphine equivalent dose

NRS Numerical Rating Scale for Pain Intensity

OC Opioid Consumption in morphine equivalent dose

OF Opioid-Free days


PACU Post Anesthesia Care Unit

PE Physical Examination

PGE Patient Global Evaluation

PK Pharmacokinetic
PT Preferred Term
QOL Quality of Life

SAE Serious Adverse Event/Experience

SAP Statistical Analysis Plan

SD Standard Deviation

SDTM Standard Data Tabulation Model

SOC System Organ Class

SRC Safety Review Committee

TEAE Treatment Emergent Adverse Event

WHO World Health Organization

WOCF Worst Observation Carried Forward


Statistical Analysis Plan Protocol Number: CA-PS-204 Date: 24APR2019

#### 1. PURPOSE OF THE ANALYSES

This statistical analysis plan (SAP) is based on protocol number CA-PS-204 Version 2.0 (28JAN2019) from Concentric Analgesics, Inc. This SAP provides details of the specific statistical methods that will be performed on data collected in this study and will be finalized and signed off before database lock.

This SAP is being written with due consideration of the recommendations outlined in the most recent International Conference on Harmonization (ICH) E9 Guideline entitled Guidance for Industry: Statistical Principles for Clinical Trials, the most recent ICH E3 Guideline and the Guidance for Industry: Structure and Content of Clinical Study and the most recent FDA draft Guidance for Industry - Analgesic Indications: Developing Drug and Biological Products, dated February 2014.

#### 2. PROTOCOL SUMMARY

#### **Study Objectives**

#### 2.1.1 Primary Objective

To evaluate the efficacy of a single intraoperative administration of CA-008 vs. vehicle placebo (100 mL volume) in subjects undergoing an elective C-ABD.

#### 2.1.2 Secondary Objective

- To evaluate the safety and tolerability of a single intraoperative administration of CA-008 vs. vehicle placebo in subjects undergoing an elective C-ABD.
- To evaluate the PK profile of a single intraoperative administration of CA-008 vs. vehicle placebo in subjects undergoing an elective C-ABD.
- To evaluate the opioid-sparing effect of CA-008 vs. placebo in subjects undergoing an elective C-ABD in terms of consumption and time to cessation.

#### 2.2 **Overall Study Design and Plan**

This is a Phase 2, single-center, randomized, double-blind, placebo-controlled, parallel design study evaluating up to 4 exploratory cohorts, each with a single dose of CA-008 or placebo.

**CONFIDENTIAL** 

For each subject, the study will be conducted in two parts:

- Inpatient period starts with admission to Post-anesthesia care unit (PACU) and continues to 96h (T96h) after completion of study treatment injection (T0).
- Outpatient period begins on discharge from the inpatient unit through various follow up visits to D29±2 (W4) after surgery, or later if necessary, for ongoing safety assessments.
   Note that additional follow up visits may occur at any time or even after D29/W4 to follow adverse events (AEs) to resolution or establishment of a new baseline.

The protocol-defined visits are presented in <u>Table 2-1</u>:

Table 2-1 Protocol-Specified Visits and Visit Windows

| Study Phase | Visit Time |
|---|---|
| Screening | From days -45 to -1 |
| Prior to Surgery/ Surgery | Day 0 |
| In-Patient (Post Surgery) | Hours 0 (post-surgery), 24, 48, 72 and 96 |
| Follow-up | Days 8(±1 day), 15(±2 days), 29(±2 days) |
| If needed, unscheduled visits or Follow Up after D29±2 | |
| Early Termination (ET) visit (for subjects who terminate early, and are agreeable to a return visit) | |

All study assessments are outlined in Table 1 of the Protocol.


# 2.2.1 Study Stopping Rules

Study enrollment will be paused if subjects experience intolerable possibly related TEAEs, as defined:

- 1 or more subjects with any grade 4 "related" TEAE in any of the categories shown in Table 2-2.
- 2 or more subjects with the same grade 3 "related" TEAE in any of the categories shown in Table 2-2.

More details are described in Section 7.2 of the Protocol.

An external independent safety review committee (SRC) will be consulted should a stopping rule be triggered to determine whether it is appropriate to continue with dosing in the study. This committee will be independent of the Sponsor or clinical research organization (CRO) and will in no way be involved with study conduct. The SRC Charter details the membership, roles and responsibilities of the SRC.


Table 2-2 Study Stopping Rules

| Category | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) | Potentially Life<br>Threatening<br>(Grade 4) |
|---|---|---|---|---|
| Abnormal Wound Healing: Infection Dehiscence Necrosis | Mild symptoms; clinical or diagnostic observations only; intervention not indicated. No interference with age-appropriate instrumental ADL | Minimal, local or<br>noninvasive<br>intervention<br>indicated; May<br>require local<br>wound care or<br>medical<br>intervention<br>(e.g., dressings<br>or topical<br>medications) | Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of existing hospitalization indicated; limiting ADLs. May require IV antibiotics, antifungals, or antivirals or radiologic intervention. | Life-threatening consequences; urgent intervention indicated |
| ECG/Cardiac<br>issues<br>Vital Signs<br>Labs | Asymptomatic, intervention not indicated | Non-urgent<br>medical<br>intervention<br>indicated | Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of existing hospitalization indicated | Life-threatening<br>consequences;<br>urgent<br>intervention<br>indicated |
| Focused Neurosensory Testing (performed by trained Investigator) | Mild symptoms | Moderate<br>symptoms;<br>limiting<br>instrumental ADL | Severe<br>symptoms<br>requiring medical<br>intervention;<br>limiting self-care<br>ADL | Life-threatening<br>and urgent<br>intervention<br>indicated |


Protocol Number: CA-PS-204 Date: 24APR2019

Statistical Analysis Plan

#### 2.2.2 Study Population

Adults ages 18 to 65 years, inclusive, who are planning to undergo an elective complete (full) abdominoplasty (C-ABD) and otherwise meet eligibility criteria may be considered for enrollment into the study.

#### 2.2.3 Treatment Regimens

Cohort #1: CA-008 5 mg vs. placebo in 100 mL of vehicle

Cohort #2: CA-008 10 mg vs. placebo in 100 mL of vehicle

Cohort #3: CA-008 15 mg vs. placebo in 100 mL of vehicle

Cohort #4 (optional): CA-008 (5mg to 15 mg) vs. placebo in 100 mL of vehicle

#### 2.2.4 Treatment Group Assignments or Randomization

Subjects who meet the enrollment criteria will be randomly allocated to receive either an active drug or placebo in a 1:1 (for Cohorts #1 or #4) or a 2 active:1 placebo ratio (for Cohorts #2 or #3). This study will use manual randomization.

Subjects who have provided written informed consent will be assigned a unique number in the screening process. This number will be used to identify the subject throughout the study. Once any subject number or randomization number is assigned, it cannot be reassigned to any other subject. Subjects may be rescreened if the screening window is exceeded due to scheduling issues.

#### 2.2.5 Sample Size Determination

There is no formal sample size estimation for this study. Given the uncertainty in estimating a sample size for C-ABD surgery, data from the current study will be used to determine the sample size for a subsequent parallel design study selecting one or more optimal doses of CA-008 vs. placebo in the setting of standard of care for abdominoplasty. The sample size is considered sufficient for that purpose.

Subjects will be randomized to either the active medication or placebo as follows:

- Cohort #1: total N=18 randomized 1:1. CA-008 5 mg or placebo
- Cohort #2: total N=18 randomized 2:1. CA-008 10 mg or placebo
- Cohort #3: total N=18 randomized 2:1. CA-008 15 mg or placebo


Protocol Number: CA-PS-204 Date: 24APR2019

Statistical Analysis Plan

• Cohort #4 (optional): total N=24 randomized 1:1 to CA-008 (5mg to 15mg) or placebo After the 3<sup>rd</sup> cohort was enrolled, the decision was made not to enroll the optional 4<sup>th</sup> cohort, therefore the final sample size will be 54 subjects.

#### 3. GENERAL ANALYSIS AND REPORTING CONVENTIONS

This section discusses general policies to be employed in the analysis and reporting of the data from the study. Departures from these general policies may be provided in the specific detailed sections of this SAP. When this situation occurs, the rules set forth in the specific section take precedence over the general policies.

Summaries and analyses will be presented separately for Cohort 1, then the other cohorts: active and placebo groups associated with Cohort 1 will be presented alone, then active arms and pooled placebo group associated with Cohorts 2, 3 and 4 (if performed) will be presented together). An overall column will be provided where appropriate.

All continuous study assessments will be summarized by treatment and time point (as applicable) using the descriptive statistics n, mean, SD, median, and range (minimum, and maximum). All categorical study assessments will be summarized by treatment and time point (as applicable) using frequency counts and rates of occurrence (%). Changes from baseline for continuous outcomes will be presented as their corresponding continuous measures for post-baseline visits if applicable. All study data will be listed by cohort, treatment, subject, and time point (as applicable).

No preliminary rounding will be performed; rounding will only occur after the analysis. To round, consider the digit to the right of the last significant digit: if <5, then round down; if ≥5, then round up. Means and medians will be presented with one more decimal place than the precision of the data. Standard deviations will be presented with two more decimal places than the precision of the data. Percentages will be presented with one decimal place. A percentage of 100% will be reported as 100%. Minimums and maximums will be presented with the same precision as the original data.

Unless otherwise indicated, all testing of statistical significance will be 2-sided, and a difference resulting in a p-value of less than or equal to 0.05 will be considered statistically significant. Furthermore, the baseline will be the last assessment before the dosing of study medication.

No adjustment will be made for multiple comparisons in this exploratory study.


Sponsor: Concentric Analgesics, Inc. Protocol Number: CA-PS-204

All analyses will be performed using the SAS System® version 9.3 or higher. For final TLFs, the domain (Study data tabulation Model [SDTM]) and analysis (Analysis Data Model [ADaM]) data sets will be taken as input to the SAS programs that generate the report-ready tables, figures and listings. The submission ready SDTM and ADaM data sets will be provided to the sponsor along with display deliveries.

Statistical Analysis Plan

Date: 24APR2019

The following conventions will be used in the study analysis as needed for intermediate calculations:

- Time 0 (T0) is the time of completion of study drug administration.
- Time P (TP) is the time of discharge from the Post anesthesia care unit (PACU)
- Day of surgery is defined as Day 0 (D0).
- Assessment visit times are defined by D0 and/or T0.
- Baseline value is defined as the last valid measurement prior to the dosing of study treatment.
- Change from baseline is defined as post-baseline value minus baseline value.
- The date/time of early termination will be the date/time that the subject confirms they no
  longer want to participate in the study, regardless of whether they decide to withdraw from
  all or only some study procedures and regardless of if they return to the site for
  assessment of wound healing.
- Duration of an AE will be computed in days for AEs lasting longer than 24 hours, and as hours for AEs lasting less than 24 hours. Duration in hours will be calculated as the stop date/time of the event minus the start date/time. Duration in days will be calculated by using stop date minus the start date +1 if AE occurs on or after taking study medication. If AE occurs prior to the study medication, then the duration will be calculated by using stop date minus the start date. If reported as ongoing at the time of database lock, the duration will be calculated using the date of the last visit or the last date of any AE for the subject in the database, whichever is later.
- The number of days in the study is computed as: [Date of study completion or withdrawal minus the date of study drug administration] + 1.


• If duplicate values are obtained at a given visit (e.g., repeated vital sign measurements), the last value will be used unless it is noted that the measurement was in error for that value. Values that compromise interpretation will not be used in summaries (e.g., values that were obtained post-dose will not be summarized as pre-dose values).

• Values that compromise interpretation will not be used in summaries (e.g., values that were obtained post-dose will not be summarized as pre-dose values).

#### 4. SUBJECT POPULATIONS

## 4.1 Analysis Populations

The following analysis populations are planned for this study:

- The Safety Population will include all subjects who received any part of a dose of study treatment.
- The PK Population will include all subjects who receive a full dose of study treatment and complete all PK assessments.
- The intent-to-treat (ITT) population will include all subjects who are randomized to study treatment.

Membership in analysis populations will be determined before unblinding.

Subjects who elect to ET after receiving study treatment and during the inpatient phase of the study will be asked to continue with assessments through T96h if they have not elected to withdraw from all aspects of study participation.

All efficacy and safety analyses will be performed using Safety population. PK analyses will be performed using PK population.

#### 4.2 Disposition of Subjects

All subjects and the populations for which they qualify will be listed. Subjects who are screened and who fail screening or withdraw consent prior to randomization or are randomized but not treated will be listed and summarized in the disposition summary table. Subjects who are randomized, subject inclusion into each study population, subjects who are treated, subjects who complete follow-up as well as subjects who withdraw early from the study and the reason for


Protocol Number: CA-PS-204 Date: 24APR2019

Statistical Analysis Plan

withdrawal will be summarized by treatment group and overall in the subject disposition summary table.

#### 4.3 Protocol Deviations

Deviations are categorized as informed consent procedures, inclusion/exclusion criteria, study medication, prohibited medications, study procedures, study drug assignment/treatment, visit or assessment time window, missed visit or assessment and/or other. All protocol deviations will be captured on case report forms (CRFs) and/or documented in site specific logs throughout the study. Deviations will be categorized and classified as major or minor by the project team and the medical monitor after database lock but before unbinding and will be discussed in the CSR. Subjects with protocol deviations, both minor and major, will be presented in a data listing and will be summarized by type of deviation and major/minor classification for all randomized subjects.

#### 5. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

#### 5.1 Demographics and Baseline Characteristics

Demographic variables include age, sex, race, and ethnicity. Baseline characteristics include height (cm), weight (kg), and body mass index (BMI; kg/m²). Demographics and baseline characteristics will be summarized overall and by treatment group using the safety population.

#### 5.2 Medical/Surgical History

Medical and Surgical history, as collected at screening, will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) version 21.0 to determine system organ class (SOC) and preferred term (PT). Medical histories will be presented in a by-subject listing. Any events that occur prior to the study procedure will be categorized as medical history.

#### 5.3 Prior and Concomitant Medications

Prior medications/therapies are those that stop prior to the start of the study drug administration. Any medication/therapy that stops at or after this time or is ongoing at the time of discontinuation/completion is considered concomitant medication/therapy. Prior and concomitant medications will be collected for the 30 days prior to screening and throughout the study. Prior and concomitant medications will be coded using World Health Organization Drug Dictionary Anatomical Therapeutic Chemical (WHO/ATC) classification index version March 1, 2018. The CONFIDENTIAL

Protocol Number: CA-PS-204 Date: 24APR2019

Statistical Analysis Plan

number and percentage of subjects who take concomitant medications will be summarized by drug class and preferred term, overall and by cohort and treatment group, for the safety population. All medications and non-medical therapies captured in CRFs will appear in data listings.

#### 6. MEASUREMENTS OF TREATMENT EXPOSURE AND COMPLIANCE

Because study medication is administered as a single dose at the study center by trained study personnel, compliance with respect to study medication will not be calculated. A listing of study drug administration and exposure data will be provided.

After completing the assessments through 96 hours after study medication administration, the diary for at-home use will be distributed to the subject to collect pain intensity (twice daily on NRS) and pain medication through Day 15. Compliance with home diary use will be evaluated based on post-discharge home diary records. Compliance for each subject will be based on the number of days the subject participated in the outpatient study period, defined as:

Where the N of expected NRS records in the diary for each subject is calculated as 2 times the number of days the subject participated in the outpatient portion of the study. The number of days of participation will be calculated as the date of the Day 15 visit or the date of the last study visit (whichever is earlier) minus the date of discharge. NRS recorded prior to a rescue use will not be included in this calculation of compliance. For example, Subject A was discharged on Day 4, if this subject discontinues the study on Day 13, then the expected N of NRS records on diary will be 18 (2 \* (13-4)). Assuming Subject A had 10 NRS available from his/her diary, then compliance for this subject would be 55.6% ((10/18) \*100). However, if subject A had discontinued the study on Day 10 (prior to Day 13), then the expected N of NRS for this subject would be 12 (2 \* (10-4)) and compliance would be 83.3% ((10/12) \*100). A summary of compliance will be provided overall, and by cohort and treatment group. Compliance with recording an NRS prior to rescue in the diary will be calculated as the number of NRS recorded prior to taking rescue medications divided by the number of rescue medication uses recorded.


#### 7. EFFICACY EVALUATION

# 7.1 Handling of Dropouts or Missing Data

All efforts will be made to minimize missing data. These efforts will include the following:

- Subjects are required to consent to continuous data collection even after discontinuation of study medication;
- Data collection will continue after subjects take rescue medication.

With the procedures above, it is expected that missing data will be minimal. Missing at random is expected to be a reasonable assumption for this study.

For the endpoints of NRS (at rest and/or after ambulation) in this study, NRS values will be imputed in the following manner:

For subjects who take rescue medication, a windowed last pain score carried forward (wLOCF) will be used. The pre-rescue pain score will be used to impute scheduled assessments for 30 minutes following the rescue use when IV fentanyl is used, 2 hours when IV hydromorphone is used, and 4 hours when PO oxycodone or other oral opioid is used.

The last NRS prior to the use of any rescue medication will be used to impute subsequent NRS at rest scores for the subsequent protocol-specified time points for measurement of pain intensity through an appropriated time window (as specified above) after the time of the dosing of the rescue medication. Note: if a pre-rescue NRS assessment occurs at the same time as a scheduled assessment, the scheduled NRS will be assumed to happen first, and then the pre-rescue NRS will be assumed to occur. If an NRS assessment occurs at the same time as the time of taking a rescue medication, the NRS will be assumed to be a Pre-rescue medication result. As an example, using PO oxycodone, if the NRS time is the same as 4 hours after taking the rescue medication (end of imputation period), then NRS will be considered as occurring before the 4 hours assessment and will be imputed. For example, if a rescue dose is taken at 1pm, all protocol-scheduled NRS will be imputed with the appropriate NRS value up to and including through 5pm. If multiple doses of rescue medication are taken within a 4-hour period, the pre-rescue NRS for the first rescue use will be carried forward continuously until 4 hours past the last use of rescue falling within the continuous window. For example, if rescue is used at Hour 2.3 and Hour 5.1, the pre-rescue NRS at Hour 2.3 will be carried forward till Hour 9.1 (5.1 +4). NRS


Statistical Analysis Plan Protocol Number: CA-PS-204 Date: 24APR2019

scores taken after ambulation will be based on reported values and the pre-rescue 4-hour imputation rule will not be used. The scores after ambulation are collected every 12 hours and no ambulation NRS score is collected prior to taking rescue medication. Intermittent missing pain scores at rest or after ambulation (due to subject sleeping, etc.) will not be imputed, and AUC will be calculated based on non-missing values. For subjects who drop out of the study, scheduled assessments will first be imputed using the worst prior pain score carried forward (WOCF). Data resulting from imputation method described above will be used in the analysis of all endpoints derived from NRS, e.g, primary endpoint (Hour 96 NRS at Rest) and key secondary efficacy endpoint (AUC<sub>(0-96)</sub> of NRS at Rest).

For categorical endpoints of PGE and IGE, assessments imputed for data after a subject discontinues from the study will be handled using a WOCF method (worst category available).

#### 7.2 **Sensitivity Analyses**

The following imputation methods will be performed and analyzed as sensitivity analyses of the primary analysis of mean NRS scores at 96 hours:

- For: subjects who drop out of the study prior to Day 15 due to Lack of Efficacy or Adverse Events, scheduled assessments to be imputed using worst prior pain score carried forward. All other subjects who drop out will have their last pain score carried forward.
- Regardless ET reasons, pain assessments after dropout to be imputed using LOCF (last scheduled non missing pain score prior to dropout
- Replace missing values after discontinuation with the within treatment median of the subjects continuing in the study.

For each of the above, values imputed after use of rescue medication will remain the same as the primary analysis.

#### 7.3 Assessment Time Windows

For calculations of all AUC endpoints and use of opioid endpoints, the actual dates/times of the assessments will be used in calculations. Thus, while the NRS are intended to be collected at the pre-defined protocol scheduled time points (e.g., Hour 0.5, 1, 2, etc.), it is recognized that operationally the scores are collected as close to the target times as possible but there is some flexibility in terms of the actual times the scores are collected. Thus, to account for this inherent


Statistical Analysis Plan Protocol Number: CA-PS-204 Date: 24APR2019

aspect of data collection, the ACTUAL TIMES will be used for the calculation of the AUC. The actual times will be based relative to the time of completion of study drug administration.

Safety assessment summaries will be based on the nominal protocol-specified assessment times.

#### 7.4 Efficacy Endpoints

## 7.4.1 Primary Efficacy Endpoint

Time-specific mean NRS pain intensity scores at T96h for CA-008 vs. placebo.

## 7.4.2 Key Secondary Efficacy Endpoints

For the CA-008 vs. placebo comparison, the following are key secondary endpoints (in descending order of importance):

- Weighted sum of pain intensity (SPI) assessments = Area Under the Curve (AUC) of the NRS current pain intensity scores from T0 to 96h at rest (AUC<sub>0 to 96h</sub>).
- Time to opioid cessation or freedom (T<sub>OF</sub>)
- Percentage of subjects who do not require opioids (i.e., opioid free; OF) from T24 to T96: OF<sub>24 to 96h</sub>
- Total opioid consumption (in daily oral morphine equivalents) = OC from T0 to T96h:  $OC_{0 \text{ to}}$ 96h

#### 7.4.3 Other Endpoints

For the CA-008 vs. placebo comparison:

- Using NRS at rest: AUC<sub>0 to 120h</sub>, AUC<sub>24 to 96h</sub>, AUC<sub>0 to W1</sub>
- AUC <sub>0</sub> to 96h (arising), AUC<sub>0</sub> to W1 (arising)
- Time-specific mean NRS scores at T48, T72, T96, T120, T144 and T168h
- OC<sub>24 to 96h</sub>
- OF<sub>24 to 96h</sub>, OF<sub>96h to W1</sub> and OF<sub>96h to W2</sub>
- The fraction of subjects who rescue at T48, T72 and T96h
- Analgesic consumption from T96h to W1 (AC<sub>96h to W1</sub>) and AC<sub>96h to W2</sub>


 PGE comparing the %age of subjects reporting "poor" + "fair" vs. "good" + "excellent" responses, and the %age reporting each category of response at T96h, D8/W1, D15/W2 and D29/W4

• IGE comparing the %age of those reporting "poor" + "fair" vs. "good" + "excellent" responses, and the %age reporting each category at T96h, D8/W1, D15/W2 and D29/W4

#### 7.5 Analysis Methods

#### 7.5.1 NRS Measurements

The NRS is an 11-point scale with anchors 0 (no pain) and 10 (worst possible pain). NRS will be assessed as follows:

- During the inpatient stay, NRS at rest beginning with the PACU admission may be assessed once the subject is awake. If the subject is able to provide responses, obtain NRS scores at T0.5, 1, 2, 4, 6, 8, 12, 16, 20, 24, and every 4 hours (if awake at time of assessment) until discharge from the inpatient unit. Time windows: for T0.5 to T2 (±5 min) and from T4 onward (±15 min).
- Pain scores may be skipped between the hours of midnight and 6 a.m., but the subject may not miss two consecutive assessments. The T12, T24, T48, T72 and T96h assessments must be completed even if the subject is asleep at these times.
- An additional NRS assessment must be obtained prior to rescue medication request (±15 min).
- During the inpatient stay, starting on postoperative day 1 (after T24) perform the following each morning at 0800h (±2h) and each evening at 2000h (±2h): document the NRS at rest and on arising. Actual assessment times must be documented. If, however these twice daily assessments coincide with timed assessments of NRS at rest, then the time assessment at rest is used in place of the twice daily assessments. Resting pain scores are performed on the schedule noted above in the first bullet.
- During the outpatient period (after T96h through W2), instruct the patient to document, if
  possible, their NRS scores twice daily at 0800h (±4h) and 2000h (±4h) at rest and on
  arising. Note that the actual time of these assessments must be documented in the diary
  whenever possible. Instruct the patient to:


 Obtain the morning NRS assessment prior to taking any pain medication or 2 (±15min) hours after taking any pain medication.

- Obtain the evening NRS assessment 2 (±15min) hours after taking any pain medication.
- 7.5.2 Time-specific mean NRS pain intensity scores at T96h (Primary Efficacy Endpoint) and other time points

Missing NRS will be handled as discussed in Section 7.1.

Mean NRS scores at specific time points will be analyzed using a 1-factor (treatment) analysis of variance (ANOVA) model with treatment as the main effect. Descriptive summaries will be presented for each treatment group. In addition, the pain intensity score at Hour 96 and at each time point will be analyzed using Wilcoxon sum-rank test for sensitivity.

7.5.3 AUC 0-96h at Rest (Key Secondary Efficacy Endpoint) and other AUC endpoints
AUC calculations will be done using the standard trapezoidal rule

AUC = 
$$\sum_{i=0}^{x} \left( \frac{NPRS_i + NPRS_{i+1}}{2} \right) * (T_{i+1} - T_i)$$

Where: NRS<sub>i</sub> = NRS at rest at time i, and  $(T_{i+1} - T_i)$  is the Time difference in hours between time i and time i+1.

Missing NRS will be handled as discussed in Section 7.1. AUC values will be analyzed using a one factor analysis of variance (ANOVA) with treatment as the main effect. Descriptive summaries (N, median, range) will be presented for each treatment group. Exact Two-Sided p-values from Wilcoxon Rank-Sum test comparing treatment group with Placebo (or Pooled Placebo) will also be presented.

Mean NRS scores (in-clinic and diary) will be graphed over time by cohort and treatment group. NRS over time by each subject may also be displayed graphically as warranted. The individual NRS and the computed AUC variables will be listed for all individual subjects.

7.5.4 Time to opioid cessation or freedom  $(T_{OF})$  (Key Secondary Efficacy Endpoint)


Protocol Number: CA-PS-204 Date: 24APR2019

Statistical Analysis Plan

Time to opioid cessation or freedom ( $T_{OF}$ ) will be defined as the time to the last use of opioid for a subject and will be analyzed using Kaplan-Meier techniques. Number of subjects with event, number of subjects censored, median time to OF, and p-values from log-rank test will be displayed in a summary table. Subjects not ceasing opioid use before ET, or until End of Study (EOS) will be censored at ET or EOS days respectively.  $T_{OF}$  starting after T24 and T48 and staying opioid free to D29 will also be derived and presented in the same table

In addition, Kaplan-Meier curves will be presented by treatment group.

7.5.5 Opioid Free (OF) 24-96h (Key Secondary Efficacy Endpoint) and other timepoints.

Opioid use is recorded on the rescue medication eCRF from the end of surgery through the D15 follow up/Early termination (ET). If additional opioids, other than the study rescue medications, appear on the concomitant medications page and can be identified, those opioids will also be considered.

The percentage of subjects who do not require opioids (are Opioid Free or OF) during each time period will be analyzed using a logistic regression or Chi Square test if there are not enough data to support the logistic regression, with treatment group as the main effect. The analysis will compare the odds ratios of the proportions of OF subjects between each treatment group and the placebo group. A summary of frequencies as well as odds ratio, 95% confidence intervals and p-values will be presented.

In addition to other specified timepoints, the proportion of subjects who are Opioid Free after T24 through D29, and the proportion of subjects who are OF after T48 through D29 will also be derived and presented.

7.5.6 Total Opioid Consumption (OC) in Daily Oral Morphine equivalents 0-96h (Key Secondary Efficacy Endpoint) and other timepoints

The amount of opioids taken as rescue will be calculated using the rescue medication page of the eCRF. If additional opioids, other than the study rescue medications, appear on the concomitant medications page and can be identified, those opioids will also be included (in terms of morphine equivalents) in the total consumed. Table 3 will be used to calculate the morphine equivalent dose (MED) for each medication. The total opioid consumption for each day for each subject will be calculated as the sum of the MEDs of all the medications taken on that day. For example, if a


subject takes 5 MED morphine on Day 1 and Day 2, and 10 MED of Oxycodone on Day 2, the total consumption for Day 1 is 5 MED, and the total consumption for Day 2 is 15 MED. Subjects that take no opioids on a day will have a total opioid consumption value of zero for that day.

 Table 3
 Equianalgesic Conversion Table

| Opioid (Doses in mg) | Conversion Factor |
|---|---|
| IV Fentanyl | 0.3 |
| PO Hydrocodone | 1 |
| PO Hydromorphone | 4 |
| PO Morphine | 1 |
| PO Oxycodone | 1.5 |
| PO Tramadol | 0.1 |
| Multiply the opioid dose by the conversion factor = oral morphine equivalent dose (MED): | |
| e.g., PO oxycodone 5 mg X 1.5 = 7.5 mg MED or | |
| IV fentanyl 25 mcg X 0. | 3 = 7.5 mg MED |

Total opioid consumption will be calculated for 0-96 hours ( $OC_{0 \text{ to } 96h}$ ) and 24-96 hrs ( $OC_{24 \text{ to } 96h}$ ). An ANOVA with treatment arm as the main effect will be performed. A separate summary containing only subjects that have taken at least one dose of rescue will be performed if warranted.

#### 7.5.7 Percentage of Subjects who Rescue at T48 and other timepoints

The percentage of subjects who rescue at T48, T72 and T96 hours will be calculated as the number of subjects who have taken at least one dose of rescue prior to the specified timepoint. The percentage of subjects who rescue during each specific time period will be analyzed using a Chi Square test. A summary of frequencies as well as odds ratio, 95% confidence intervals and p-values will be presented. (OC)

#### 7.5.8 PGE and IGE

The proportions of subjects in each individual PGE or IGE category will be summarized by treatment group and analyzed using the Cochran-Mantel-Haenszel (CMH) mean score test (using equally spaced scores) at each time point they are collected to compare treatments across the 4 levels of outcomes (poor, fair, good, or excellent). In addition, Fisher's exact test will be performed to compare treatments across 2 levels of outcomes (Poor/Fair versus Good/excellent).


Statistical Analysis Plan Sponsor: Concentric Analgesics, Inc. Protocol Number: CA-PS-204

Individual PGE and IGE scores will be listed.

#### 8. SAFETY EVALUATION

#### 8.1 **Overview of Safety Analysis Methods**

All safety outcomes will be summarized using the safety population. No formal statistical comparisons will be performed for safety outcomes. Safety outcomes include:

 Incidence of spontaneous reported treatment-emergent adverse events (TEAEs) or serious adverse events (SAEs)

Date: 24APR2019

- Physical examination (PE)
- Vital signs
- Surgical site assessments
- Neurosensory testing near the incision
- Rebound or worsening pain
- ECG
- Clinical laboratory test results

#### 8.2 Adverse Events and SAEs

All AEs will be listed, but only TEAEs will be summarized.

Treatment-emergent AEs are defined as any of the following:

- Non-serious AEs with onset on the date of treatment with the study drug through Day 29 or Early Termination, whichever occurs first.
- Serious AEs with onset on the date of treatment with the study drug through 30 days after Day 29 or Early Termination, whichever occurs first.
- AEs that start before the start of treatment but increase in severity or relationship at the time of or following the start of treatment through Day 29 or Early Termination, whichever occurs first.

For evaluation of causal relatedness to treatment, the categories are probably related, possibly related or unlikely related. For categorization in the summary tables, AEs designated as probably or possibly related will be considered related.


Statistical Analysis Plan Protocol Number: CA-PS-204 Date: 24APR2019

For the evaluation of event severity terms, the criteria are mild, moderate, severe or potentially life-threatening. In addition to a listing of all TEAEs, treatment related TEAEs, serious TEAEs, Deaths, and TEAEs leading to premature discontinuation from the study will be provided.

An overall summary will be prepared giving for each treatment group and overall, both the number of TEAEs, and the number of subjects with at least one TEAEs, as well as SAEs, treatment related TEAEs and TEAEs leading to premature discontinuation from study.

The number of subjects with AEs will be summarized for each treatment group and overall by SOC and PT sorted in alphabetically by SOC, and then by PT within SOC. These summaries will be given by cohort and treatment in separate tables for each of the following TEAE event sets:

- All events
- Treatment related events
- Serious events
- Events leading to premature discontinuation from study
- Events by maximum severity
- Events by Relationship to Study Drug

If a given subject experiences a TEAE that maps to the same PT/SOC more than once, the subject will be counted only once for the SOC/PT at the greatest severity (i.e., mild, moderate, or severe) and causality (i.e., related).

Duration of a TEAE lasting more than 24 hours will be computed in days as the stop date of the event minus the start date plus 1 and will be reported in days. TEAEs lasting less than 24 hours will be computed as stop date/time minus start date/time and reported in hours. If reported as ongoing at the time of database lock, the stop date is defined as the date of the last visit or the last date of any event for the subject in the database, whichever is later.

If a TEAE is considered resolved, but the stop date is missing, the last day of the month will be imputed if the month and year are available. If only the year is available, and the year is the same as the year of the last visit, the stop date will be the latest of the last visit date or latest event for the subject in the database.

If the year of the event is prior to the year of the last treatment, the end day and month will be set to 31 December.

 Sponsor: Concentric Analgesics, Inc. Protocol Number: CA-PS-204

For missing or partial start and stop dates/times, the most conservative imputation will be used (AEs will be assumed to be temporally related to the study medication). <u>Table 4</u> will be used to impute any missing dates/times:

Statistical Analysis Plan

Date: 24APR2019


Table 4 Table of Imputation Rules for Missing AE Start Dates

| Missing Date<br>Portion | Prior to<br>Treatment | Same as Treatment<br>Start Date | After Treatment Start<br>Date |
|---|---|---|---|
| Day | Month and Year <<br>Month and Year of<br>Study treatment: | Month and Year =<br>Month and Year of<br>Study treatment: | Month and Year ><br>Month and Year of<br>Study Treatment: |
| | Start Day = 1 | Start Day = Day of first<br>treatment | Start Day = 1 |
| | Stop Day=last day of the month | Stop Day= last day of the month | Stop Day=last day of the month |
| Day and Month Define Day as | Year < Year of first treatment: | Year = Year of study treatment: | Year > Year of study<br>treatment: |
| above, then: | Start Month = July | Start Month = Month of<br>study treatment | Start Month = January |
| | Stop Month = Dec | Stop Month = Dec | Stop Month = Dec |
| Day, Month, and<br>Year | | | |
| Time | Missing start times will be imputed as 00:01 | | |
| | Missing stop times will be | e imputed as 23:59 | |

After following these imputation rules, if the start date/time is imputed as a date after the end date/time, the start date/time will be set to the end date/time to provide a positive duration for the event incidence.

Missing assessments for AE study medication relationship or severity will be analyzed as related or severe respectively. No other imputation is planned for safety data.

#### 8.3 Physical Examination

A complete medical history and physical examination including all major body systems will be performed at Screening. In addition, a focused interim medical history and targeted physical examination will be performed prior to surgery (if not done on D-1), and to capture changes after


Protocol Number: CA-PS-204 Date: 24APR2019

Statistical Analysis Plan

Surgery, at 96 hours (± 4 hours) after the administration of study medication, but prior to discharge, and Days 8, 15 and 29/ET after the administration of study medication.

Abnormal or clinically significant physical exam will be recorded as AEs. Physical examination results will be listed for individual subjects.

#### 8.4 Vital Signs

Vital signs results including blood pressure (systolic and diastolic; mmHg), heart rate (beats per minute), respiration rate (breaths/min), and temperature will be listed for individual subjects.

Baseline for vital signs measurements will be defined as the last evaluation before dosing with study medication. Summary statistics, including change from baseline, will be determined for each measure and will be summarized by treatment and time point.

#### 8.5 Surgical Site Assessments and Rebound (or Worsening) Pain Assessments

Surgical sites will be assessed at 48 hours (±2 hours) and 96 hours (±4 hours after study medication administration but prior to discharge from the inpatient unit) and then as an outpatient on Days 8, 15 and 29. The investigator will evaluate their satisfaction with the healing of the wound during this surgical site assessment using an 11-point scale (0- 10) where a score of 0 is "completely unsatisfied" and a score of 10 is "completely satisfied). In addition, subjects will report whether they have noted any worsening pain (rebound pain; Y/N) at the surgical site since the prior visit at Days 8, 15 and/or 29.

All data will be presented in data listings. Results of surgical site assessments and the number of subjects with rebound pain will be summarized descriptively by treatment and time point.

#### 8.6 Neurosensory Test

Neurosensory testing of the area proximal to the surgical incision approximately 3 cm from the incision will be performed at Screening visit, 48 hours (±2 hours), 96 hours (±4 hours, but prior to discharge) and Day 8, Day 15 and Day 29 after the administration of study medication or if the subject terminates early, at that time if allowed.

The neurosensory assessment results will be listed and the number of subjects in each response will be summarized descriptively by treatment group and time point for each wound (cephalad or caudad).


Protocol Number: CA-PS-204 Date: 24APR2019

Statistical Analysis Plan

#### 8.7 ECG

ECG examination will be assessed at screening and 24 hours (±2 hours) after study medication administration.

Number of subjects with abnormal results will be summarized by treatment and time point. All ECG data will be listed.

#### 8.8 Clinical Laboratory Test Results

Clinical laboratory tests (chemistry, hematology, coagulation and urinalysis) will be collected at screening and before discharge from the inpatient unit (T96h). All results will be listed. For each lab test, the raw value and change from screening will be summarized by treatment group.

Each clinical laboratory test will be defined by the clinical laboratory to be "Low", "Normal", or "High", according to the normal reference range from the clinical laboratory.

The number and percentage of subjects who have a shift from within to outside the normal reference range from screening to T96h will be summarized for overall, and by cohort and treatment.

## 8.9 Drugs of Abuse and Alcohol Screens, Pregnancy Test

Pregnancy (for female subjects of childbearing potential), urine drug screen and alcohol (breath or saliva) tests will be performed at screening and pre-surgery.

Results will be listed for individual subjects. Each test result will be defined to be "negative" or "positive".

#### 8.10 Subject Pain Assessment Training and Surgery Details

Pain assessment training will be provided during screening. Subjects will re-watch video prior to surgery. Patient pain assessment training and surgery details will be documented in CRFs and will be listed for each subject.

#### 9. PHARMACOKINETIC EVALUATION

The time points for PK whole blood collections will be at baseline (from Check-in and up to 30 min prior to surgery), 5, 10, 15, 30, 45 minutes, and at hours 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 30, 36 and 48 (for a total of 20 samples) after the end of study treatment administration.


Actual sampling times will be used to calculate plasma-derived PK parameters. Full details of PK endpoints/analyses will be described in a separate PK Analysis plan.

#### 10. OTHER ANALYSES

N/A

#### 11. INTERIM ANALYSES

N/A

#### 12. REFERENCES

US Federal Register. (1998) International Conference on Harmonization; Guidance for Industry: Statistical Principles for Clinical Trials. Department of Health and Human Services: Food and Drug Administration. Federal Register, Vol. 63, No. 179, September 16, 1998, page 49583.

US Federal Register. (1996) International Conference on Harmonization; Guidance for Industry: Structure and Content of Clinical Study Reports. Department of Health and Human Services: Food and Drug Administration. Federal Register Vol. 61, July 17, 1996, page 37320.

Guidance for Industry (2014) Analgesic Indications: Developing Drug and Biological Products - Draft Guidance. Department of Health and Human Services: Food and Drug Administration. Center for Drug Evaluation and Research (CDER) February 2014 Clinical/Medical.

#### 13. APPENDICES

#### 13.1 Planned Tables, Figures and Listings

# 13.1.1 Tables

| Table 14.1.1 | All Subjects | Summary of Subject Disposition |
|---|---|---|
| Table 14.1.2 | Randomized | Summary of Protocol Deviations |
| | Subjects | |
| Table 14.1.3 | Safety | Summary of Demographics and Baseline Characteristics |
| | Population | |
| Table 14.1.4 | Safety | Summary of Concomitant Medications by ATC Class and |
| | Population | Preferred Term |
| Table 14.1.5 | Safety | Summary of Subject NRS and NRS at Rescue Diary Compliance |
| | Population | |
| Table 14.2.1.1 | Safety | ANOVA Analysis of Hour 96 NRS at Rest – WOCF (Primary Analysis) |
| | Population | |


| T 44.0.4.0 | | |
|---|---|---|
| Table 14.2.1.2 | Safety | Wilcoxon Analysis of Hour 96 NRS at Rest – WOCF (Sensitivity |
| Table 44 0 4 0 | Population | Analysis) |
| Table 14.2.1.3 | Safety<br>Population | ANOVA Analysis of Hour 96 NRS at Rest – WOCF and LOCF (Sensitivity Analysis) |
| Table 14.2.1.4 | Safety | ANOVA Analysis of Hour 96 NRS at Rest – LOCF (Sensitivity |
| 14510 11.2.1.1 | Population | Analysis) |
| Table 14.2.1.5 | Safety | ANOVA Analysis of Hour 96 NRS at Rest – Median (Sensitivity |
| | Population | Analysis) |
| Table 14.2.2.1 | Safety | ANOVA Analysis of NRS at Rest by Hour |
| | Population | |
| Table 14.2.2.2 | Safety<br>Population | ANOVA Analysis of NRS at Rest by Morning/Night |
| Table 14.2.2.3 | Safety | Wilcoxon Analysis of NRS at Rest by Hour |
| | Population | , |
| Table 14.2.2.4 | Safety | Wilcoxon Analysis of NRS at Rest by Morning/Night |
| | Population | |
| Table 14.2.3.1 | Safety | ANOVA Analysis of AUC (0-96) NRS at Rest – WOCF (Key |
| | Population | Secondary Efficacy Analysis) |
| Table 14.2.3.2 | Safety | Wilcoxon Analysis of AUC (0-96) NRS at Rest – WOCF |
| | Population | |
| Table 14.2.3.3 | Safety | ANOVA Analysis of AUC over Various Time Periods NRS at Rest – |
| | Population | WOCF |
| Table 14.2.3.4 | Safety | ANOVA Analysis of AUC over Various Time Periods upon Arising - |
| | Population | WOCF |
| Table 14.2.4 | Safety | Log-Rank Analysis of Time to opioid cessation or freedom (ToF) (Key |
| | Population | Secondary Efficacy Analysis) |
| Table 14.2.5 | Safety | Logistic Analysis of Proportion of Subjects Who Are Opioid Free at |
| | Population | Various Time Periods (Key and Exploratory Secondary Efficacy |
| | | Analysis) |
| Table 14.2.6 | Safety | Logistic Analysis of Proportion of Subjects Who Rescue at Various |
| | Population | Time Periods |
| Table 14.2.7 | Safety | ANOVA Analysis of Opioid Consumption (in Morphine Equivalents) |
| | Population | (Key Secondary and Exploratory Efficacy Analysis) |
| Table 14.2.8 | Safety | CMH Analysis of Patient Global Evaluation at T96h and Other Time |
| | Population | Periods |
| Table 14.2.9 | Safety | CMH Analysis of Investigator Global Evaluation at T96h and Other |
| | Population | Time Periods |
| Table 14.3.1 | Safety | Overall Summary of Treatment-Emergent Adverse Events (TEAEs) |
| | Population | _ ` , |
| Table 14.3.1.1 | Safety | Summary of Treatment-Emergent Adverse Events (TEAEs) by System |
| | Population | organ Class and Preferred Term |
| Table 14.3.1.2 | Safety | Summary of Treatment Related Treatment-Emergent Adverse Events |
| | Population | (TEAEs) by System organ Class and Preferred Term |
| Table 14.3.1.3 | Safety | Summary of Serious Adverse Events by System organ Class and |
| | Population | Preferred Term |
| Table 14.3.1.4 | Safety | Summary of Treatment-Emergent Adverse Events (TEAEs) Leading to |
| | Population | Study Discontinuation by System organ Class and Preferred Term |
| | opalation | , |


| Table 14.3.1.5 | Safety | Summary of Treatment-Emergent Adverse Events (TEAEs) by System organ Class, Preferred Term and Severity |
|---|---|---|
| Table 14.3.1.6 | Population<br>Safety | Summary of Treatment-Emergent Adverse Events (TEAEs) by System |
| 1 4 5 1 1 1 5 1 1 5 | Population | organ Class, Preferred Term and Relationship to Study Drug |
| Table 14.3.2.1 | Safety | Summary of Chemistry Laboratory Tests: Results and Change from |
| | Population | Baseline |
| Table 14.3.2.2 | Safety<br>Population | Summary of Chemistry Laboratory Tests: Shift from Baseline |
| Table 14.3.3.1 | Safety | Summary of Coagulation Laboratory Tests: Results and Change from |
| | Population | Baseline |
| Table 14.3.3.2 | Safety | Summary of Coagulation Laboratory Tests: Shift from Baseline |
| | Population | |
| Table 14.3.4.1 | Safety | Summary of Hematology Laboratory Tests: Results and Change from |
| | Population | Baseline |
| Table 14.3.4.2 | Safety | Summary of Hematology Laboratory Tests: Shift from Baseline |
| | Population | |
| Table 14.3.5.1 | Safety | Summary of Urinalysis Laboratory Tests: Results and Change from |
| | Population | Baseline |
| Table 14.3.5.2 | Safety | Summary of Urinalysis Laboratory Tests: Shift from Baseline |
| | Population | |
| Table 14.3.6 | Safety | Summary of Vital Signs: Results and Change from Baseline |
| | Population | |
| Table 14.3.7 | Safety | Summary of Surgical Site Assessment |
| | Population | |
| Table 14.3.8 | Safety | Summary of Rebound Pain Assessment |
| | Population | |
| Table 14.3.9.1 | Safety | Summary of Neurosensory Exam – Cephalad to Wound |
| | Population | |
| Table 14.3.9.2 | Safety | Summary of Neurosensory Exam – Caudad to Wound |
| | Population | |
| Table 14.3.10 | Safety | Summary of ECG Exam Abnormal Findings |
| | Population | |


# 13.1.2 Figures

| Figure 14.2.1 | Safety Population | Mean NRS scores over time (in-clinic and diary) by Treatment Group |
|---|---|---|
| Figure 14.2.2 | Safety Population | NRS over time for each subject by Cohort |


# 13.1.3 Listings

| | I | I = |
|---|---|---|
| Listing 16.2.1 | All Subjects | Randomization and Study Population |
| Listing 16.2.2 | All Subjects | Informed Consent and Re-Consent |
| Listing 16.2.3 | All Subjects | Eligibility |
| Listing 16.2.4 | All Subjects | Protocol Deviations |
| Listing 16.2.5 | All Subjects | Subject disposition/ Early Termination |
| Listing 16.2.6 | All Randomized Subjects | Demographics and Baseline Characteristics |
| Listing 16.2.7 | All Randomized Subjects | Medical/ Surgical History |
| Listing 16.2.8.1 | All Randomized Subjects | Prior and Concomitant Medications |
| Listing 16.2.8.2 | All Randomized Subjects | Rescue Medication Administration |
| Listing 16.2.8.3 | All Randomized Subjects | Non-Medication Therapies |
| Listing 16.2.9 | All Randomized Subjects | Surgery |
| Listing 16.2.10 | All Randomized Subjects | Study Drug Administration, Pain Assessment Training and Discharge |
| Listing 16.2.11 | All Randomized Subjects | Subject NRS and NRS at Rescue Diary Compliance |
| Listing 16.2.12.1 | All Randomized Subjects | Pain Intensity Assessment (NRS at Rest) |
| Listing 16.2.12.2 | All Randomized Subjects | Pain Intensity Assessment (NRS on Arising) |
| Listing 16.2.13 | All Randomized Subjects | List of Efficacy Endpoints |
| Listing 16.2.14 | All Randomized Subjects | Patient Global Evaluation (PGE) |
| Listing 16.2.15 | All Randomized Subjects | Investigator Global Evaluation (IGE) |
| Listing 16.2.16.1 | All Randomized Subjects | Adverse Events |
| Listing 16.2.16.2 | All Randomized Subjects | Serious Adverse Events |
| Listing 16.2.16.3 | All Randomized Subjects | Treatment Related Adverse Events |
| Listing 16.2.16.4 | All Randomized Subjects | Adverse Events Leading to Study Discontinuation |
| Listing 16.2.17.1 | All Randomized Subjects | Chemistry Laboratory Test Results |
| Listing 16.2.17.2 | All Randomized Subjects | Coagulation Laboratory Test Results |
| Listing 16.2.17.3 | All Randomized Subjects | Hematology Laboratory Test Results |
| Listing 16.2.17.4 | All Randomized Subjects | Urinalysis Laboratory Test Results |
| Listing 16.2.18 | All Randomized Subjects | Vital Signs |
| Listing 16.2.19 | All Randomized Subjects | Alcohol Breath and Urine Drug Screen Tests |
| Listing 16.2.20 | All Randomized Subjects | Pregnancy Test |
| Listing 16.2.21 | All Randomized Subjects | Physical Examination and Targeted Physical Exam |
| _ | | Assessment |
| Listing 16.2.22 | All Randomized Subjects | Surgical Site Assessment and Rebound Pain |
| 11.41.42.22.2 | | Assessment |
| Listing 16.2.23 | All Randomized Subjects | Neurosensory Exam |
| Listing 16.2.24 | All Randomized Subjects | 12-Lead Electrocardiogram |
| Listing 16.2.25 | PK Population | Pharmacokinetic (PK) Concentration Data |


# **14. DOCUMENT HISTORY**

| Version<br># | Summary of Changes | Section Changed | Date |
|--------------|---------------------------|-----------------|-----------|
| 1.0 | Initial document released | NA | 24Apr2019 |

